CLINICAL TRIAL: NCT00389480
Title: A Phase I Study of DB-67 (7-t-butyldimethylsilyl-10-hydroxycamptothecin) in Adult Patients With Refractory or Metastatic Solid Malignancies
Brief Title: Study of AR-67 (Formerly DB-67) in Adult Patients With Refractory or Metastatic Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arno Therapeutics (Industry)
Collaborators: University of Kentucky (Other); Arch Medical Services Inc., DBA The Center for Cancer Care and Research (Industry)
Responsible Party: Arno Therapeutics, Arno Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARN-AR67-CT101
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Tumors
Keywords: Solid Tumors; Solid Malignancies; Phase I
MeSH Terms: conditions — Neoplasms | interventions — 7-tert-butyldimethylsilyl-10-hydroxycamptothecin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Dose escalating
  Interventions: Drug: AR-67 (formerly DB-67)

INTERVENTIONS:
Drug: AR-67 (formerly DB-67) — infusion daily x 5 days, every 21 days

SUMMARY:
Hypothesis:

AR-67 (formerly DB-67) represents a rationally engineered drug that possesses improved stability, toxicity, and efficacy compared to current Food and Drug Administration (FDA)-approved camptothecins, based on the extensive research of prior studies. Therefore, the investigators hypothesize that AR-67 (formerly DB-67) will be well-tolerated and efficacious in phase I clinical trials. This initial phase I trial will establish the maximum tolerated dose in humans, establish the toxicity profile, and define the appropriate dose of AR-67 (formerly DB-67) for future phase II and III clinical trials.

DETAILED DESCRIPTION:
Overview of Study:

Camptothecins are a potent class of anticancer drugs that inhibit DNA topoisomerase I. Topotecan and irinotecan are two FDA approved second generation congeners currently in clinical use, and have a spectrum of activity which includes colorectal, ovarian, and lung cancers. Unfortunately, these drugs are hampered by a labile α-hydroxy-δ-lactone pharmacophore, which hydrolyzes to yield the inactive carboxylate form of the drug.

AR-67 (formerly DB-67) (7-t-butyldimethylsilyl-10-hydroxycamptothecin) is a third generation analog engineered to be blood stable and highly potent. Its enhanced stability results from two factors: (1) AR-67 (formerly DB-67) is highly lipophilic, partitioning into lipid bilayers, thus protecting it from hydrolysis in the aqueous milieu of the bloodstream, and (2) the 10-hydroxy functionality of the drug effectively ablates the high affinity interactions of the carboxylate drug form with albumin, which has been previously shown to diminish the levels of the active lactone species in the circulation.

On the basis of its stability and activity, AR-67 (formerly DB-67) was selected by the National Cancer Institute (NCI) for development in the first cycle of the Rapid Access to Intervention Development (RAID) program. Data from cycle I, as well as independent data from collaborative efforts, revealed impressive in vitro and in vivo antitumor activity, particularly in an intracranial glioma model system. Through the continued support of the RAID program, the drug has been extensively studied in mice, rats and beagle dogs and the pre-clinical MTD has been determined. After extensive investigation of various formulations, a Cremophor:ethanol compound has been identified as the most appropriate for the phase I study in humans and the GMP grade drug product has been refined and completed. This protocol describes the initial phase I study in humans using AR-67 (formerly DB-67).

Primary Endpoint:

* To estimate the MTD and describe the DLT of intravenous AR-67 (formerly DB-67) administered once daily for 5 days every 21 days to adults with recurrent or refractory solid tumors in which standard therapies are not effective.

Secondary Endpoints:

* To characterize the plasma pharmacokinetics of AR-67 (formerly DB-67) and its metabolites after intravenous administration.
* To explore the pharmacogenetic effects of polymorphisms in drug metabolism and transport mediated by liver enzymes and by efflux or uptake proteins, respectively, and relate these polymorphisms to AR-67 (formerly DB-67) pharmacokinetics and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* >18 year old subjects with solid malignancies that have progressed after at least one prior chemotherapy regimen and have exhausted other therapies
* Treated and clinically stable brain metastases
* Measurable OR non-measurable disease
* Greater than three weeks since surgery
* Normal organ and marrow function
* ECOG Performance Status of < 2
* No other prior malignancy except for treated basal cell or squamous cell skin cancer, in situ cervical cancer, Stage I or II cancer (patient in complete remission) or other cancer from which the patient has been disease-free for 5 years.
* Computed tomography (CT) scan of involved areas within 28 days of registration
* Life expectancy of greater than 12 weeks.

Exclusion Criteria:

* Pregnant or nursing females
* Chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) of entering the study.
* Patients may not be receiving any other investigational agent. Uncontrolled intercurrent illness including active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Allergic reactions to compounds of similar chemical or biologic composition to DB-67 (i.e. camptothecins such as irinotecan, topotecan, or others of this class of pharmaceuticals).
* Subjects with prior anaphylactic injection reaction of > grade 3 to paclitaxel or any other product formulated with cremophor
* Subjects with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Any time during the four 21-day cycles
Dose limiting toxicity (DLT) | Any time during the four 21-day cycles

SECONDARY OUTCOMES:
Pharmacokinetics | at each dose during week 1
Pharmacogenetic effects of polymorphisms | at each dose during week 1

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Arch Medical Services Inc. DBA The Center for Cancer Care and Research, St Louis, Missouri